CLINICAL TRIAL: NCT00662376
Title: Safety, Tolerance and Metabolic Effects of Using a Preoperative Oral Nutritional Supplement (PreOP Booster) in Gastrointestinal Surgery
Brief Title: Study on Safety, Tolerance and Metabolic Effects of a Nutritional Supplement, Given as a Drink Before Gallbladder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Dr. Steffen Benzing, Kabi Innovation Centre, Fresenius Kabi Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-POB-01-UK
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-11

CONDITIONS: Enteral Nutrition Regimen Prior to Surgery
MeSH Terms: interventions — Dietary Supplements; Food

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Test (Experimental): oral nutritional supplement (assignment: according to consecutive random numbers)
  Interventions: Dietary Supplement: PreOP Booster (oral nutritional supplement, food for special medical purposes)
- Control (Placebo Comparator): placebo (assignment: according to consecutive random numbers)
  Interventions: Dietary Supplement: PreOP Booster (oral nutritional supplement, food for special medical purposes)

INTERVENTIONS:
Dietary Supplement: PreOP Booster (oral nutritional supplement, food for special medical purposes) — 3 x 1 dosages of oral nutritional supplement / placebo are given prior to surgery: 2 the evening before the day of operation and 1 dosage 3-4 h before initiation of anaesthesia

SUMMARY:
The aim of this pilot study is to obtain data on the safety, tolerance and metabolic effects of the oral nutritional supplement (PreOP Booster) given to patients prior to gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy

Exclusion Criteria:

* bile duct stones
* ileus
* conditions affecting gastric emptying
* severe, organ-specific disorders
* HIV
* inherited metabolic disorders
* known intolerance against or allergy to any component of the investigational feeds

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety parameters reflecting pathophysiological functions of the liver | day -1, 0, 1, and 7
Gastrointestinal tolerance | day 0 before and 6-8h after surgery
Metabolic parameters in serum, liver and muscle tissue | on day -1, 0, 1, and 7

SECONDARY OUTCOMES:
Clinical parameters (infectious and non-infectious complications) | until day 7

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N. Lobo, MS, DM, FRCS, Principal Investigator — Queen's Medical Centre, Division of Gastrointestinal Surgery, Nottingham University Hospitals;
Locations (1):
- Queen's Medical Centre, Division of Gastrointestinal Surgery, Nottingham University Hospitals;, Nottingham, United Kingdom

REFERENCES:
- [Derived] Awad S, Stephens F, Shannon C, Lobo DN. Perioperative perturbations in carnitine metabolism are attenuated by preoperative carbohydrate treatment: Another mechanism by which preoperative feeding may attenuate development of postoperative insulin resistance. Clin Nutr. 2012 Oct;31(5):717-20. doi: 10.1016/j.clnu.2012.02.015. Epub 2012 Mar 22. PMID 22444237
- [Derived] Awad S, Constantin-Teodosiu D, Constantin D, Rowlands BJ, Fearon KC, Macdonald IA, Lobo DN. Cellular mechanisms underlying the protective effects of preoperative feeding: a randomized study investigating muscle and liver glycogen content, mitochondrial function, gene and protein expression. Ann Surg. 2010 Aug;252(2):247-53. doi: 10.1097/SLA.0b013e3181e8fbe6. PMID 20622656